CLINICAL TRIAL: NCT06023173
Title: Deep Radiomics-based Fusion Model Predicting Bevacizumab Treatment Response and Outcome in Patients With Colorectal Liver Metastases: a Multicenter Cohort Study
Brief Title: Deep Radiomics-based Fusion Model Predicting Bevacizumab Treatment Response and Outcome in Patients With Colorectal Liver Metastases
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Head of Colorectal Surgery, Fudan University
Other Study IDs: DERBY
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: The Patients With CRLM Who Benefit More From Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Training Cohort: This cohort was derived from Arm A (treated with FOLFOX + bevacizumab) of the BECOME studyand was used for model construction.
  Interventions: Diagnostic Test: Deep radiomics-based fusion model
- Negative Validation Cohort: The cohort was derived from Arm B (treated with FOLFOX) of the BECOME study , which demonstrated that the model specifically predicted the efficacy of bevacizumab.
  Interventions: Diagnostic Test: Deep radiomics-based fusion model
- Internal Validation Cohort: The cohort was derived from an independent Zhongshan Hospital cohort with the same treatment team and imaging instrumentation as the BECOME study, differing only in patient period, and was used for internal validation of the model.
  Interventions: Diagnostic Test: Deep radiomics-based fusion model
- External Validation Cohort: The cohort was obtained from the Zhongshan Hospital - Xiamenand the First Affiliated Hospital of Wenzhou Medical University for external validation of the model.
  Interventions: Diagnostic Test: Deep radiomics-based fusion model

INTERVENTIONS:
Diagnostic Test: Deep radiomics-based fusion model — This multi-modal deep radiomics model, using PET/CT, clinical and histopathological data, was able to identify patients with bevacizumab-sensitive CRLM, providing a favorable approach for precise patient treatment.
  Other Names: deep learning model

SUMMARY:
This multi-modal deep radiomics model, using PET/CT, clinical and histopathological data, was able to identify patients with bevacizumab-sensitive unresectable colorectal cancer liver metastases, providing a favorable approach for precise patient treatment.

DETAILED DESCRIPTION:
Accurately predicting tumor response to targeted therapies is essential for guiding personalized conversion therapy in patients with unresectable colorectal cancer liver metastases (CRLM). Currently, tumor response evaluation criteria are based on assessments made after at least 2-months treatment. Consequently, there is a compelling need to develop baseline tools that can be used to guide therapy selection. Herein, the investigators proposed a deep radiomics-based fusion model which demonstrates high accuracy in predicting the efficacy of bevacizumab in CRLM patients. Further, the investigators observed a significant and positive association between the predicted-responders and longer progression-free survival as well as longer overall survival in CRLM patients treated with bevacizumab. Moreover, the model exhibits high negative prediction value, indicating its potential to accurately identify individuals who are unresponsive to bevacizumab. Thus, our model provides a valuable baseline method for specifically identifying bevacizumab-sensitive CRLM patients, which is offering a clinically convenient approach to guide precise patient treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤75 years;
2. Patients were histologically confirmed for colorectal adenocarcinoma with unresectable liver-limited or liver-dominant metastases
3. PET/CT at baseline were available
4. First line treated with FOLFOX+ bevacizumab.

Exclusion Criteria:

1. Resectable liver metastases;
2. Wide-type KRAS/NRAS;
3. No measurable liver metastasis;
4. No efficacy assessment;
5. No follow-up information.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this multicenter cohort study, the investigators collected 307 patients with colorectal cancer liver metastases. The training cohort and negative validation cohort were derived from the BECOME study (NCT01972490), for whom baseline PET/CT images were available. The internal validation cohort was derived from consecutive metastastic colorectal cancer patients of the multi-disciplinary team (MDT) at Zhongshan Hospital (ZSH), share the same MDT, surgical team, and PET/CT imaging equipment with training cohort, from 01 January 2018 to 31 December 2018. The external validation cohort came from the MDT of Zhongshan Hospital - Xiamen and the First Hospital of Wenzhou Medical University, from 01 January 2020 to 31 December 2020
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
ORR | 2013.10.1-2023.1.1
  Objective response rate of patients with colorectal cancer liver metastases who treated with FOLFOX+bevacizumab/FOLFOX
PFS | 2013.10.1-2023.1.1
  Progression-free survival of patients with colorectal cancer liver metastases who treated with FOLFOX+bevacizumab/FOLFOX

SECONDARY OUTCOMES:
OS | 2013.10.1-2023.1.1
  Overall survival of patients with colorectal cancer liver metastases who treated with FOLFOX+bevacizumab/FOLFOX

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, MD, Principal Investigator — Fudan University
Locations (1):
- Department of General Surgery, Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No